CLINICAL TRIAL: NCT05765461
Title: Effect of Lipikar Baume AP+M on Quality of Life and Pain Related to Atopic Dermatitis and Other Skin Diseases With Dryness or Severe Xerosis on Adults
Brief Title: Effect of Lipikar Baume AP+M on Quality of Life and Pain of Adults With Dryness or Severe Xerosis
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP20001-LIPIKAR BAUME AP+M
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis; Skin Diseases
Keywords: atopic dermatitis; severe xerosis; quality of life; dryness
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at evaluating the effect of a topical product on the improvement of quality of life and pain of patients suffering from atopic dermatitis or other skin diseases with dryness or severe xerosis. Patients aged 16 years and over are asked to apply the product once or twice a day for 2 months. They may be prescribed a corticosteroid upon decision of the dermatologist.

DETAILED DESCRIPTION:
The general approach of the statistical methodology is the following:

* The qualitative variables are described with number and percent of each level.
* The quantitative variables are described with mean and standard deviation.
* All statistical hypotheses are performed at the 5% significance level using 2-sided tests.
* Given the large sample size, no normality assessment will be done.
* Mean reduction rate for quantitative variables is calculated as (mean v0 - mean v1)/mean v0)*100.
* Due to the high number of zeros at inclusion in the self-assessment quantitative criteria, analyses will concern only patient with an intensity above 0 at inclusion or at final visit.
* Response rate for qualitative variables is calculated as the percent of patients with at least on level decrease between the two visits.
* Response rate for satisfaction is the percent of patients declaring being Satisfied or Very satisfied.
* Response rate for tolerance is the percent of patients declaring the tolerance High or Excellent.

ELIGIBILITY:
Inclusion Criteria:

• atopic dermatitis or other skin disease with dryness or severe xerosis

Exclusion Criteria:

• patients not suffering from atopic dermatitis or other skin disease with dryness or severe xerosis

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients meeting the inclusion criteria and agreeing to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 4631 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
change in the intensity of skin disease | from baseline to Day56
  The dermatologist evaluates the intensity of the skin condition on a 5-point scale (from absent to very severe)

SECONDARY OUTCOMES:
change in the intensity of skin dryness | from baseline to Day56
  The dermatologist evaluates the intensity of the skin condition on a 5-point scale (from absent to very severe)
evolution of the inflammatory lesions surface | from baseline to Day56
  The dermatologist evaluates the inflammatory lesions surface with the following scale:
  * none
  * <10%
  * [10%;30%[
  * >30%
change in the intensity of pruritus | from baseline to Day56
  The dermatologist evaluates the intensity of pruritus on a 5-point scale (from absent to very severe)
change in the quality of sleep | from baseline to Day56
  The dermatologist evaluates the intensity of pruritus on a 5-point scale (from unaffected to very severely affected)
change in the daily discomfort | from baseline to Day56
  The dermatologist evaluates the intensity of the daily discomfort on a 5-point scale (from absent to very severe)

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Kerob, Study Director — Cosmetique Active International
Locations (7):
- Dermatology practices, Zagreb, Croatia
- Dermatology practices, Berlin, Germany
- Dermatology practices, Lisbon, Portugal
- Dermatology practices, Pretoria, South Africa
- Dermatology practices, Taipei, Taiwan
- Dermatology practices, Bangkok, Thailand
- Dermatology practices, Hanoi, Vietnam